CLINICAL TRIAL: NCT04443569
Title: Lidocaine Patches After Cesarean Section
Acronym: LPACS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2000028500
Record Dates: First submitted 2020-06-19; First posted 2020-06-23 (Actual); Results first posted 2023-10-10 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-10

CONDITIONS: Postoperative Pain; Obstetric Pain; Opioid Use
MeSH Terms: conditions — Pain, Postoperative; Labor Pain

STUDY DESIGN:
Intervention Model Description: This will be a prospective randomized non-blinded controlled trial. All cesarean sections for women undergoing their first or second cesarean delivery will be included. Patients will be approached and consented during the pre-operative period when presenting for scheduled surgery or at the time of consent for a non-scheduled cesarean section. The lidocaine patch would be placed on the superior-lateral aspect of the Pfannenstiel incision in the PACU prior to being transferred to the postpartum floor.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor/statistician will not be made aware of the treatment group of the patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lidocaine Patch Group (Experimental): This group will be women who were randomized to receive a lidocaine patch for postoperative pain following cesarean delivery in addition to routine postoperative pain management.
  Interventions: Drug: Lidocaine patch
- Control Group (Placebo Comparator): This group will be women randomized to routine postoperative pain management following cesarean delivery. A placebo patch will be placed superior to the Pfannenstiel incision in the same manner as the lidocaine patch treatment group.
  Interventions: Other: Placebo patch

INTERVENTIONS:
Drug: Lidocaine patch — Lidocaine patch to be placed in post-operative recovery area and used in addition to routine post-cesarean delivery pain management
  Arms: Lidocaine Patch Group
Other: Placebo patch — A placebo patch will be placed superior to the Pfannenstiel incision in the same manner as the lidocaine patch treatment group.
  Arms: Control Group

SUMMARY:
The aim of this study is to investigate the impact of using lidocaine patches after cesarean section on pain control and opioid use in the immediate post-operative period. The hypothesis is the use of lidocaine patches in the immediate post-operative period will lead to a decrease in the visual analog pain score compared to women who do not use a lidocaine patch in the immediate post-operative period following cesarean delivery. Additionally, a decrease in the use of opioids as pain control compared to patients that do not have a lidocaine patch in place the is anticipated.

DETAILED DESCRIPTION:
The use of lidocaine as a local anesthetic is a common and widely used in practice. Lidocaine patches can be used for localized pain control and can be placed every 24 hours. The use of lidocaine patches in post-operative patients has been reported in one case report in obstetric literature. There is one study that reports decreased immediate postoperative pain when lidocaine patches were placed at laparoscopic port sites following gynecologic surgery as measured by visual analog scale score and the Prince Henry and 5-point verbal rating pain scale. There have been no studies looking at the impact of lidocaine patches in obstetric surgical procedures, specifically cesarean sections.

Cesarean sections are one of the most common surgeries in the United States. Following cesarean sections it is common to utilize opioids in the hospital and upon discharge to manage patient's post-operative pain. According to the CDC overdose deaths involving prescription opioids were five times higher in 2017 than in 1999 with over 200,000 deaths. This creates an opportunity to decrease the use of post-operative opioids with the application of a lidocaine patch as an adjunctive post-operative pain management modality following cesarean sections.

Lidocaine patches are a common topical analgesia therapy used for localized pain control in the inpatient and outpatient setting. It's use in the postoperative period is less understood and the use of topical lidocaine patches has not been thoroughly investigated in the surgical literature. Thus far, it has been shown as an effective therapy at laparoscopic port sites following laparoscopic appendectomies. It's use in obstetrical surgeries has not been studied. Overall, the limited research on this topic making it a valuable area of research.

This study will involve prospective enrollment of women undergoing cesarean deliveries. Women will be randomized to receive a lidocaine patch or no lidocaine patch to be worn for 72 hours after delivery to help manage postoperative pain. This will be an adjunctive therapy in addition to the parental and oral narcotic pain medication that is routine prescribed. The utility of lidocaine patches for management of post-cesarean delivery pain will be assess by 2 measures. The first measure will involve the total daily dose of narcotic used in morphine equivalent doses. The second outcome assessed will be subjective pain as measured on a 1-10 scale and reported by the patients to nursing staff. This score will be averaged for each 24 hour period post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Primary or secondary cesarean delivery
* Able to consent to research study

Exclusion Criteria:

* 3 or more prior cesarean deliveries
* History of abdominoplasty
* History of abdominal hernia repair with mesh
* Allergy to lidocaine
* Allergy to adhesives in medical tape
* Women who received general anesthesia for their cesarean delivery
* Women with active substance abuse
* Women methadone or suboxone for a history of opiate abuse

Ages: 18 Years to 52 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Patients need to be pregnant and undergoing a cesarean delivery
Enrollment: 93 (Actual)
Dates: Start 2021-10-10 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Audrey Merriam, MD, MS, Principal Investigator — Assistant Professor; Assistant Professor, Department of Obstetrics, Gynecology and Reproductive Sciences; Christopher Arkfeld, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gilhooly D, McGarvey B, O'Mahony H, O'Connor TC. Topical lidocaine patch 5% for acute postoperative pain control. BMJ Case Rep. 2011 Feb 8;2011:bcr0620103074. doi: 10.1136/bcr.06.2010.3074. PMID 22715181
- [Background] Kwon YS, Kim JB, Jung HJ, Koo YJ, Lee IH, Im KT, Woo JS, Im KS. Treatment for postoperative wound pain in gynecologic laparoscopic surgery: topical lidocaine patches. J Laparoendosc Adv Surg Tech A. 2012 Sep;22(7):668-73. doi: 10.1089/lap.2011.0440. Epub 2012 Aug 3. PMID 22861076
- See also: Related Info — https://casereports.bmj.com/content/2011/bcr.06.2010.3074

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lidocaine Patch Group | Control Group
Started | 46 | 47
Completed | 46 | 47
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lidocaine Patch Group | Control Group | Total
Number analyzed (Participants) | 46 | 47 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.4 (3.9) | 33.5 (4.6) | 33.4 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 47 | 93
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 13 | 25
  Not Hispanic or Latino | 34 | 34 | 68
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 6 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 5 | 13
  White | 27 | 33 | 60
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 3 | 11
Region of Enrollment [Number; unit: participants]
  United States | 46 | 47 | 93
Prepregnancy Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 30.4 (7.8) | 29.6 (6.6) | 30 (7.2)
BMI at Delivery [Mean (Standard Deviation); unit: kg/m^2] | 35.3 (6.9) | 34.5 (6.7) | 34.9 (6.8)
Gravidity [Mean (Standard Deviation); unit: pregnancies] — The number of times a woman has been pregnant, regardless of whether the pregnancies were interrupted or resulted in a live birth.
  pregnancies | 3.2 (1.6) | 3.4 (2) | 3.3 (1.8)
Parity Term [Mean (Standard Deviation); unit: births] — Number of births a female has had after 20 weeks gestation.
  births | 1.3 (0.8) | 1.5 (0.9) | 1.4 (0.8)
Parity Preterm [Mean (Standard Deviation); unit: births] — Number of births a female has had before 20 weeks gestation.
  births | 0.2 (1.3) | 0.1 (0.3) | 0.2 (1.0)
Parity Abortions [Mean (Standard Deviation); unit: births] — Number of births a female has had resulting in abortions.
  births | 0.9 (1.5) | 0.9 (1.2) | 0.9 (1.3)
Parity Living Children [Mean (Standard Deviation); unit: births] — Number of births a female has had resulting in living children.
  births | 1.4 (0.9) | 1.6 (0.9) | 1.5 (0.9)
Gestational Age at Delivery [Mean (Standard Deviation); unit: weeks] | 38.6 (1) | 38.4 (1.3) | 38.5 (1.2)
Number of Previous C-sections [Mean (Standard Deviation); unit: c-sections] | 1 (0.7) | 1.1 (0.7) | 1.1 (0.7)

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Pain Score
Description: Daily pain scores conducted by the nursing staff every morning and prior to medication administration. This will be a repeated measure using the subjective 0-10 pain scale. The scores will be averaged over each 24 hour (day) period and then compared. Lower scores indicate less pain.
Time Frame: the first 72 hours post-operative, up to 4 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lidocaine Patch Group | Control Group
Number analyzed (Participants) | 46 | 47
score on a scale
  Post-Op Day 1 | 3.5 (2.3) | 4.1 (2.5)
  Post-Op Day 2 | 5.2 (2.6) | 5.2 (2)
  Post-Op Day 3 | 5.2 (2.1) | 4.3 (1.7)
  Post-Op Day 4 | 5.7 (1.9) | 4.5 (2.1)
Statistical Analysis 1: Comparison: Lidocaine Patch Group vs Control Group; Post-Op Day 1; Test type: Superiority; p = 0.3, t-test, 2 sided
Statistical Analysis 2: Comparison: Lidocaine Patch Group vs Control Group; Post-Op Day 2; Test type: Superiority; p = 0.9, t-test, 2 sided
Statistical Analysis 3: Comparison: Lidocaine Patch Group vs Control Group; Post-Op Day 3; Test type: Superiority; p = 0.07, t-test, 2 sided
Statistical Analysis 4: Comparison: Lidocaine Patch Group vs Control Group; Post-Op Day 4; Test type: Superiority; p = 0.09, t-test, 2 sided

2. Secondary Outcome: Narcotic Use
Description: The total average milligrams of narcotic, or opioid, medication that a patient receives calculated in morphine equivalents
Time Frame: the first 72 hours post-operative
Measure: Mean (Standard Deviation); unit: mg morphine equivalents
Arm/Group | Lidocaine Patch Group | Control Group
Number analyzed (Participants) | 46 | 47
mg morphine equivalents | 51.3 (53.6) | 29.7 (35)
Statistical Analysis 1: Comparison: Lidocaine Patch Group vs Control Group; Test type: Superiority; p = 0.02, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: the first 72 hours post-operative
Groups:
- Control Group: This group will be women randomized to routine postoperative pain management following cesarean delivery.
Arm/Group | Lidocaine Patch Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/47
Other Adverse Events (participants affected / at risk) | 0/46 | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-24): https://cdn.clinicaltrials.gov/large-docs/69/NCT04443569/Prot_SAP_000.pdf